CLINICAL TRIAL: NCT02285426
Title: A Multicenter Study Evaluating the Diagnostic Value for Vascular Abnormalities of High Definition Bronchoscopy When Combined With I-scan Imaging Technology Compared to High Defintion Bronchoscopy Alone
Brief Title: HD+ I-scan Bronchoscopy Vascular Abnormalities Detection Multicenter Study
Acronym: i-scan
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL5012109114
Record Dates: First submitted 2014-10-27; First posted 2014-11-07 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Lungcancer
Keywords: i-scan; histology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — biopsy of sites with abnormal or suspicious vascular patterns
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- suspected lungcancer: Patients will undergo a bronchoscopy with the Pentax EB1990i HD-bronchoscope investigating the entire bronchial tree. The HD+ bronchoscopy needs to be performed in a standardized way using 3 different imaging modes:
  1. HD+bronchoscopy
  2. HD+bronchoscopy + i-Scan 1
  3. HD+bronchoscopy + i-Scan 2
  Interventions: Device: Pentax EB-1990i HD-bronchoscope guided biopsy

INTERVENTIONS:
Device: Pentax EB-1990i HD-bronchoscope guided biopsy — 3 different types of bronchoscopy image settings will be used investigating the entire bronchial tree.
  When sites with abnormal or suspicious vascular patterns are detected meeting the criteria of abnormality [visual scale adapted from Herth 2009 and Zaric 2013] the investigator will change to a normal bronchoscope and take biopsies from each site and a biopsy from a normal secondary carina on the contralateral site as control.

SUMMARY:
Videobronchoscopy is an essential diagnostic procedure for evaluation of the central airways and pivotal for the diagnosis and staging of lung cancer. Further technological improvements have resulted in high definition (HD+) images and advanced image enhancement technique (i-scan). An earlier study (NCT01676012) has indicated that HD+ bronchoscopy in combination with i-scan technology is superior to HD+WL (white light) for detecting endobronchial vascular changes. In this study we aim to correlate these vascular changes to histology and hypothesize that these vascular changes are related to (pre-) malignant changes and that the addition of i-scan is superior to HD+ WL.

DETAILED DESCRIPTION:
Patients will undergo a bronchoscopy with Pentax EB1990i HD-bronchoscope in combination with Pentax EPKi series videoprocessor investigating the entire bronchial tree. Bronchoscopy will be performed by an experienced chest physician under local anaesthesia use and type of sedation following local protocol. Bronchoscopy will be performed in a standardized order using three different imaging modes. The order of the different modes will be randomized to avoid induced scope and / or cough lesion bias. High definition digital videos will be made from all procedures without in screen patient identification, but using a study code. The three imaging modes used in this study are: HD+, HD+ surface enhancement (SE, i-scan1) and HD+ surface enhancement and tone enhancement (TE-c, i-scan2).

When sites with abnormal or suspicious vascular patterns are detected the investigator grade these findings using a visual classification scale [adapted from Herth JTO 2009 & Zaric Med Oncol 2013] and change to a regular bronchoscope and take biopsies from each site and a biopsy from a normal secondary carina on the contralateral site as control. Finally any other indicated procedures will be performed at the discretion of the local investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for diagnostic bronchoscopy for suspected or proven lung cancer.
* ASA physical status 1-3.
* Age 18 years or older.
* Signed and dated patient informed consent.

Exclusion Criteria:

* Bleeding disorders.
* Indication for use of anticoagulant therapy (acenocoumarol, warfarin, therapeutic dose of low molecular weight heparines or clopidrogel).
* Known allergy for lidocaine.
* Known pulmonary hypertension.
* Recent and/or uncontrolled cardiac disease.
* Compromised upper airway (eg concomitant head and neck cancer or central airway stenosis for any reason).
* ASA classification greater than or equal to 4.
* Pregnancy.
* Inability to consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or proven lung cancer are eligible if there is an indication for bronchoscopy. Eligible are patients with ASA physical status 1-3 and aged 18 years or older.
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
positive predictive value of HD+ i-scan bronchoscopy for detecting (pre-) malignant lesions | 7 days
  Determing the positive predictive value of HD+ i-scan bronchoscopy for vascular pattern detection .

SECONDARY OUTCOMES:
correlation between endobronchial vascular patterns and histology | 7 days
  relate grading of detected vascular abnormalities with histology outcome of biopsies
interobserver variability for detecting vascular abnormalities | 3 - 12 months
  compare bronchoscopist reported outcome to central review of obtained videos to determine interobserver variability
impact of HD-bronchoscopy on clinical decision | 1-56 days
  interview based evaluation to investigate whether the use of of i-scan technology and or the outcome of study-detected vascular sites changed the clinical approach or follow-up plan

CONTACTS AND LOCATIONS:
Overall Officials: Erik HF van der Heijden, MD, PhD, Principal Investigator — Principal Investigator
Locations (4):
- Ospedale Umberto I, Via Dante Alighieri n.1, Ravenna, RA, Italy
- RadboudUMC, Nijmegen, Gelderland, Netherlands
- St-Petersburg Research Institute of TB and Thoracic Surgery, Saint Petersburg, Russia
- Hospital Universitario Santa Lucia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Heijden EHFM, Candoli P, Vasilev I, Messi A, Perez Pallares J, Yablonskii P, van der Vorm A, Schuurbiers OCJ, Hoefsloot W. Image enhancement technology in bronchoscopy: a prospective multicentre study in lung cancer. BMJ Open Respir Res. 2018 May 18;5(1):e000295. doi: 10.1136/bmjresp-2018-000295. eCollection 2018. PMID 29862031